CLINICAL TRIAL: NCT00804661
Title: Predictors of Nocturnal Hypoventilation in Patients With Cystic Fibrosis
Brief Title: Sleep in Patients With Cystic Fibrosis
Acronym: Sommeil
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Yannick Vacher, Department Clinical Research of Developpement
Other Study IDs: P070202
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-05

CONDITIONS: Cystic Fibrosis
Keywords: sleep; nocturnal hypoventilation; sleep quality; lung function
MeSH Terms: conditions — Cystic Fibrosis; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children and adults with cystic fibrosis
  Interventions: Device: SENTEC device

INTERVENTIONS:
Device: SENTEC device — Nocturnal recording SAO2 and PtcCO2 and wrist movements by means of actigraphy
  Other Names: Nocturnal SAO2/PtcCO2 and wrist movements

SUMMARY:
The aim of the study is to identify the parameters that are associated with nocturnal hypoventilation in children and adults with cystic fibrosis. Included patients will undergo a nocturnal evaluation of their gas exchange and sleep quality by actigraphy during their annual check up. The aim is thus to identify which parameters (such as lung function parameters) are associated with nocturnal hypercapnia or hypoxemia and/or poor sleep quality

DETAILED DESCRIPTION:
Background In patients with cystic fibrosis (CF), respiratory disease is characterised by a progressive and ineluctable decline in lung function. Sleep-disordered breathing may occur at an early stage of lung disease and may impair quality of life. Oxygen therapy or noninvasive positive pressure ventilation may improve nocturnal hypoxemia and hypercapnia.Risk factors for nocturnal hypercapnia or hypoxemia are not well identified in patients with CF.

Type of study : prospective, transversal, open

Methods :

During the annual check up, a sleep study will be performed with a nocturnal recording of a least 6 hours of pulse oximetry (SaO2) and transcutaneous carbon dioxide (PtcCO2) by the SENTEC device and wrist movements by means of actigraphy. The results of the sleep study will be correlated to·

* clinical scores which evaluate sleep quality (such as the PITTSBURG Sleep Quality Score).·
* respiratory function parameters : lung volumes, forced expiratory of the respiratory muscles: maximal inspiratory and expiratory pressures and the sniff nasal inspiratory pressure.·
* nutritional state with the body mass index z-score·
* the presence of arterial pulmonary hypertension on an echocardiography·
* infectious status (colonisation by Staphylococcus aureus or Pseudomonas aeruginosa) and the CFTR genotype.

Expected results This study should be able to document abnormal nocturnal gas exchange and sleep-disordered breathing in patients with CF in a stable state. The identification of parameters associated with nocturnal hypoventilation and/or poor sleep quality will help to screen those patients who will need a sleep study and treatment such as oxygen therapy or noninvasive positive pressure ventilation.

ELIGIBILITY:
Inclusion Criteria:

* children > 8 years and adults with CF
* in a stable state (no acute respiratory exacerbation since one month or patient finishing an antibiotic course)
* able to perform reproducible forced expiratory flows
* having a forced expiratory volume in one second ≤ 60% predicted value
* who accepts to perform a sleep study in the hospital during one night
* written agreement to participate to the study

Exclusion Criteria:

* acute respiratory exacerbation in the previous month or patient who has not finished an antibiotic course
* Inability or impossibility to perform reproducible forced expiratory flows (pneumothorax during the previous year and/or without surgery)
* having a forced expiratory volume in one second > 60% predicted value
* refusal or impossibility to perform a sleep study in the hospital during one night
* patients receiving long term oxygen therapy or noninvasive positive pressure ventilation
* no social security
* impossibility of a medical examination

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the pneumology centers participating to the study
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine clinical and functional parameters associated with nocturnal hypoventilation defined by· - A mean transcutaneous carbon dioxide pressure (PtcCO2) ≥ 45 mm Hg· - And/or a maximal PtcCO2 ≥ 55 mm Hg· - And/or a PtcCO2 ≥ 45 mm Hg during ≥ 50% | At the inclusion visit

SECONDARY OUTCOMES:
To determine clinical and functional parameters associated with- sleep -disordered breathing defined by the presence of arousals on actigraphy (Actiwatch™) in children and adults with CF - nocturnal hypoxemia defined by -- a mean pulse oximetry (SaO2) | At the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Fauroux, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- AP-HP, Armand Trousseau hospital, Paris, France